CLINICAL TRIAL: NCT00249249
Title: Study of Pitavastatin 2 mg vs. Atorvastatin 10 mg and Pitavastatin 4 mg vs. Atorvastatin 20 mg (Following Up Titration) in Patients With Primary Hypercholesterolemia or Combined Dyslipidemia
Brief Title: Study to Compare the Efficacy of Pitavastatin With That of Atorvastatin in Lowering Cholesterol Levels
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kowa Research Europe (Industry)
Responsible Party: Neil Hounslow, MD, Kowa Research Europe, Ltd.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NK-104-301; EudraCT number 2005-001000-39
Record Dates: First submitted 2005-11-04; First posted 2005-11-07 (Estimated); Results first posted 2009-12-16 (Estimated); Last update posted 2010-01-12 (Estimated); Status verified 2010-01

CONDITIONS: Primary Hypercholesterolemia; Dyslipidemia
Keywords: hypercholesterolemia; dyslipidemia; kowa; KRE; pitavastatin; NK-104
MeSH Terms: conditions — Dyslipidemias; Hypercholesterolemia | interventions — pitavastatin; Atorvastatin

INTERVENTIONS:
Drug: Pitavastatin
Drug: Atorvastatin

SUMMARY:
The purpose of this study is to compare the efficacy of pitavastatin with that of atorvastatin.

DETAILED DESCRIPTION:
Following a wash-out dietary lead-in period, patients will receive either Atorvastatin or Pitavastatin during 12 weeks, in order to establish the efficacy of pitavastatin in reducing cholesterol levels.

ELIGIBILITY:
Inclusion Criteria:

* Males and females (age 18-75 years).
* Non-pregnant, non-lactating females
* Women of child bearing potential should use sustained contraceptive preparations or an approved mechanical contraceptive method.
* Eligible and able to participate and have given informed consent
* Must have been following a restrictive diet and does not eat or drink grapefruit
* Diagnosis of primary hypercholesterolemia or combined dyslipidemia
* Available for every clinic visit, which will occur in the morning.

Exclusion Criteria:

* Homozygous familial hypercholesterolemia or familial hypoalphalipoproteinemia
* Conditions which may cause secondary dyslipidemia.
* Condition which might significantly alter the absorption, distribution, metabolism, or excretion of any drug.
* History of pancreatic injury or pancreatitis, or impaired pancreatic function/injury
* Liver injury
* Impaired renal function
* Current obstruction of the urinary tract or difficulty in voiding due to mechanical as well as inflammatory conditions, which is likely to require intervention during the course of the study or is regarded as clinically meaningful by the investigator
* Serum creatine kinase (CK) >5 x upper limit of the reference range (ULRR).
* Uncontrolled hypothyroidism
* Severe acute illness or severe trauma in the last 3 months
* Major surgery, 3 months prior to Visit 1
* Significant cardiovascular disease (CVD) prior to randomization
* Evidence of symptomatic heart failure, gross cardiac enlargement; significant heart block or cardiac arrhythmias. History of uncontrolled complex ventricular arrhythmias, uncontrolled atrial fibrillation/flutter or uncontrolled supraventricular tachycardias with a ventricular response rate of >100 beats per minute at rest.
* Left ventricular (LV) ejection fraction < 0.25
* History of symptomatic cerebrovascular disease
* Conditions at the discretion of the investigator
* Known HIV infection
* Poorly controlled or uncontrolled hypertension.
* Known muscular or neuromuscular disease of any type
* Neoplastic disease
* Drug abuse or continuous consumption of more than 65 mL pure alcohol per day
* Exposure to any investigational new drug within 30 days of study entry or ingestion of any drug known to be toxic to a major organ system
* Current or recent use of supplements known to alter lipid metabolism
* Hypersensitivity reactions to other HMG-CoA reductase inhibitors
* Concomitant medication not permitted
* Resistant to lipid-lowering medications. Known hypersensitivity or intolerance to any lipid lowering agent
* Excessive obesity
* Regular clinic attendance in the morning impractical
* Signs of mental dysfunction or other factors likely to limit ability to cooperate

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 830 (Actual)
Dates: Start 2005-10; Study Completion 2006-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dragos Budinski, Med Dr., Study Director — Kowa Research Europe
Locations (192):
- Denmark (6):
  - Copenhagen University Hospital, Copenhagen
  - Medical Center, Copenhagen
  - Y Forskning, Bispebjerg Hospital, Copenhagen Nv
  - Frederiks Hospital, Kardiologisk, Frederiksberg
  - Kolesterollaboratoriet, Hellerup
  - CCBR A/S, Vejle
- Finland (5):
  - Geri-Med Oy, Helsinki
  - Kaisaniemen Laakariasema, Helsinki
  - keravan Laakarikeskus, Helsinki
  - SOK-tyoterveyshuolto, Tampere
  - TYKS University Hospital, Turku
- Germany (20):
  - Kardiologische Gemeinschaftspraxis Prof. Reifart, Bad Soden/Taunus
  - Praxis Dr. Boenninghoff, Beckum
  - Klinische Forschung Berlin Mitte, Berlin
  - Gemeinschaftspraxis am Bahnhof, Berlin-Spandau
  - Pharmakologisches Studienzentum Chemnitz, Chemnitz
  - GWT-TUK mbH, Zentrum fur Klinische Studien, Dresden
  - Internistische Diabetische Schwerpunktpraxis Dr., Frankfurt am Main
  - Gemeinschaftspraxis Dr. Krause, Th. Menke, Goch
  - Klinische Forschung Hamburg, Hamburg
  - Innere Medizin I/Medizinische Klinik, Heidelberg
  - Gemeinschaftspraxis H. Holz Dr. Med, K. W. Klingl, Lampertheim
  - ZET-Studien GmbH Leipzig, Leipzig
  - Internistische Gemeinschaftspraxis, Mainz
  - Praxis Dr. Wachter, Mannheim
  - Gemeinschaftspraxis Melcherstaette, Melcherstaette
  - Gemeinschaftspraxis Dr. Senftleber, Dr. Kohler, Messkirch
  - Praxisgemeinschaft im Kleinen Biergrund, Offenbach/M
  - Gemeinschaftspraxis Drs. Mockesch, Weinheim
  - Intermed Institud Fur Klinische Forschung und Arzn, Wiesbaden
  - Gemeinschaftspraxis Dr. Emden, Frank Drewes, Worpswede
- India (21):
  - Apollo Hospital, Andhra Pradesh
  - Care Hospital, Andhra Pradesh
  - School of Diabetology, Nizam Institute of Medical Sciences, Andhra Pradesh
  - Bhagwan Mahaveer Jain Heart Centre, Bangalore
  - Sri Ramachandra Medical College Hospital, Chennai
  - Heart Care Clinic, Gujarat
  - Apollo Hospitals, Hyderabaad
  - CARE Group of Hospitals, Hyderabaad
  - St. John's Medical College Hospital,, Karnataka
  - St. John's Medical College Hospital, Karnataka
  - Bathia Hospital, Maharashtra
  - LTMMC & General Hospital, Maharashtra
  - Sir J. J. Group of Hospitals, Maharashtra
  - King Edward Medical College & Hospital, Maharashtra
  - Ruby Hall Clinic, Maharashtra
  - Lokmanya Hospital, Maharashtra
  - PD Hinduja Hospital, Mumbai
  - Apollo Hospital, New Delhi
  - Sir Gagaram Hospital, New Delhi
  - Apollo Hospital, Tamil Nadu
  - Department of Cardiology, Tamil Nadu
- Israel (9):
  - Department of Internal Medicine, Soroka Medical Center, Beersheva
  - Department of Internal Medicine A, Rambam Medical Center, Haifa
  - Department of Internal Medicine, Wolfson Medical Center, Holon
  - Center for Research, Hadassah University Hospital, Jerusalem Ein Kerem
  - Meir Hospital, Kfar Saba
  - Department of Medicine, Hadassah Medical Center, Mount Scopus Jerusalem
  - Department of Internal Medicine, Rivka Sieff Medical Center, Safed
  - Institute of Metabolic Diseases, Tel Aviv
  - Institute of Lipid & Atherosclerosis Research, Tel Litwinsky
- Italy (10):
  - Dipartimento di Medicina Clinica e Biotecnologia Applicata, Bologna
  - Centro di Ricerca Clinica, Chieti
  - Gerontologia e Geriatria - Universita degli Studi, Ferrara
  - Dipartimento di Medicina Interna DIMI, Genova
  - Universita di Modena e Reggio Emilia, Policlinico, Modena
  - Dipartimento di Medicina Clinica e Sperimentale, Napoli
  - Medicina Clinica e delle Patologie Emergenti, Palermo
  - Dipartimento di Medicina Interna e Scienze Biomediche, Parma
  - U.O Malattie Metaboliche e Diabetologia, Treviglio
  - Azienda Ospedaliero-Universitaria, Trieste
- Netherlands (19):
  - Andromed Breda, Breda
  - Middellaan 5, Breda
  - Andromed Eindhoven, Eindhoven
  - Bomanshof 8, Eindhoven
  - Andromed Noord, Groningen
  - Damsterdiep 9, Groningen
  - Vasculair Onderzoek Centrum Hoorn, Hoorn
  - Andromed Leiden, Leiden
  - Doezastraat 1, Leiden
  - Andromed Nijmegen, Nijmegen
  - Kamerlingh Onnesstraat 16-18, Nijmegen
  - Andromed Rotterdam, Rotterdam
  - Mathenesserlaan 247, Rotterdam
  - Albert Schweitzer Ziekenhuis, Sliedrecht
  - Andromed Oost, Velp
  - Reigerstraat 30, Velp
  - Rivierenland Tiel, Wp Tiel
  - Andromed Zoetermeer, Zoetermeer
  - Parkdreef 142, Zoetermeer
- Norway (5):
  - Volvat Medisinske Senter, Fredrikstad
  - Nyomen Legekontor, Kongsberg
  - Radhuset Spesialistsenter, Oslo
  - Rikshospitalet - University Hospital, Oslo
  - Skedsmo Medisinske Senter A.S., Skedsmokorset
- Poland (10):
  - Podlaski Osrodek Kardiologii, Bialystok
  - NZOZ GCP Dobra Praktyka Lekaska, Gruziadz
  - NZOZ Terapia Optima, Katowice
  - NZOZ Centrum, Poradnia Kardiologiczna, Siedlce
  - Spec. Gab. Lek. Internistyczno-Kardiologicznly, Tarnów
  - Woj.Szp.Spec.Nr 1 im. Prof. J. Gasinskiego, Tychy
  - Instytut Zywnosci i Zywienia, Warsaw
  - Lecznica PROSEN SMO, Warsaw
  - Szpital Wolski im. Dr A. Gostynskiej, Warsaw
  - NZOZ Esculap, Przychodnia Lekary Rodzinnych, Łosice
- Russia (28):
  - Kemerovo Cardiology Dispensary, Kemerovo
  - Central Clinical Hospital 1 of RZD, Moscow
  - City Clinical Hospital 23, Moscow
  - City Clinical Hospital 64, Moscow
  - Federal State Institution Out-Patient Clinic ï€£3 of Russian Federation of Presidentâ€™s Management, Moscow
  - Federal State Institution Outpatient Clinic ï€£3 of Russian Federation of Presidentâ€™s Management, Moscow
  - Moscow City Clinical Hospital 68, Moscow
  - Moscow Regional Research Clinic Institute n.a.M.F.Vladimirov, Department of Therapy, Moscow
  - State Educational Institution of Higher Professional Education â€œMoscow State University of Medicine and Dentistry of Federal Agency of Health Care and Social Developmentâ€�, Department of Internal Diseases and Rheumatology based at City Clinica, Moscow
  - State Educational Institution of Higher Professional Education â€œMoscow State University of Medicine and Dentistry of Federal Agency of Health Care and Social Developmentâ€�, Hospital Therapy Department # 1 based at City Clinical Hospital # 40, Moscow
  - State Educational Institution of Higher Professional Education â€œMoscow State University of Medicine and Dentistry of Federal Agency of Health Care and Social Developmentâ€�, Hospital Therapy Department #1 based at City Clinical Hospital # 52, Moscow
  - State Educational Institution of Higher Professional Education â€œRussian State Medical University Federal Agency of Health Care and Social Developmentâ€�, Department of Polyclinic Therapy based at Diagnostic Center # 1, Moscow
  - State Educational Institution of Higher Professional Education â€œRussian State Medical University Federal Agency of Health Care and Social Developmentâ€�, Department of Therapy based at City Hospital # 4, Moscow
  - State Educational Institution of Higher Professional Education â€œRussian State Medical University of Federal Agency of Health Care and Social Developmentâ€�, Department of Hospital Therapy #1 based at City Clinical Hospital #15, Cardiology Dept, Moscow
  - State Institution â€œResearch Institute of Physical and Chemical Medicineâ€� of Federal Agency of Health Care and Social Development, Laboratory of Clinical Cardiology based at Bauman City Hospital # 29, Moscow
  - State Institution â€œRussian Cardiology Research Complexâ€� of Federal Agency of Health Care and Social Development, Myasnikov Clinical Cardiology Institute, Department of Hemodialysis and Plasmapheresis, Moscow
  - State Research Center for Preventive Medicine, Moscow
  - Novosibirsk Reg. Clinical Cardiology Dispensary, Novosibirsk
  - Central Medical Unit 122, St. Pb, Saint Petersburg
  - Clinical Hospital of Russian Academy of Sciences, Saint Petersburg
  - Consulting and Diagnostic Center 85, Saint Petersburg
  - Krestovsky Island Medical Institute, Saint Petersburg
  - Pokrovskaya City Hospital, Saint Petersburg
  - St. Petersburg State Medical Institution â€œOut-patient Clinic # 109â€�, Saint Petersburg
  - St. Petersburg State Medical Institution â€œOutpatient Clinic # 109â€�, Saint Petersburg
  - St. Petersburg State Medical Institution â€œPokrovskaya City Hospitalâ€�, Cardiology Department #2, Saint Petersburg
  - State Educational Institution of Higher Professional Education, â€œSaint-Petersburg State Medical University n.a.Academician I.P.Pavlov of Federal Agency of Health Care and Social Developmentâ€�, Chair and Department of Faculty Therapy, Saint Petersburg
  - State Educational Institution of Higher Professional Education, â€œSaint-Petersburg State Medical University n.a.Academician I.P.Pavlov of Federal Agency of Health Care and Social Developmentâ€�, Institute of Cardiovascular Diseases, Saint Petersburg
- Spain (19):
  - Hospital Clinico S. Juan de Alicante, San Juan, Alicante
  - Hospital Clinic i Provincial, Villaroel, Barcelona
  - Hospital de San Vicente, Alicante
  - Hospital Santa Creu I Sant Pau,, Barcelona
  - Hospital Santa Creu I Sant Pau, Barcelona
  - Hospital Universitario de Bellvitge, Barcelona
  - Hospital Vall d'Hebron, Barcelona
  - Hospital Universitario Reina Sofia, Córdoba
  - Hospital Ramon y Cajal, Madrid
  - Centro de Especialidades Pedro Gonzalez Bueno, Madrid
  - Fundacion Jimenez Diaz, Madrid
  - Hospital Clinico San Carlos, Madrid
  - Centro de Salud de Ventanielles, Oviedo
  - Hospital Marques de Valdecilla, Santander
  - Hospital Clinico Universitario de Santiago, Santiago de Compostela
  - Hospital Virgen del Roci-o, Seville
  - Hospital Dr. Peset, Valencia
  - Hospital Clinico Lozano Blesa, Zaragoza
  - Hospital Miguel Servet, Zaragoza
- Sweden (10):
  - Angelholms Sjukhus, Medicinkliniken, Angelhom
  - Sahlgrenska University Hospital, Intermedicin, Gothenburg
  - Hjartmottagningen, Helsingborg
  - Lakarcentrum Nyponet, Karineholm
  - Medicinkliniken, Ludvika
  - Huslakaren i Sandviken, Sandviken
  - Narsjukhuset Sandviken, Kardiologlab, Medicin, Sandviken
  - Hjart & Karlcenter, Södertälje
  - Karolinska Universitetssjukhuset, Stockholm
  - Hjarthuset AB, Varberg
- United Kingdom (30):
  - Oldfield Surgery, Bath
  - St James's Surgery, Bath
  - St Michael's Partnership, Bath
  - The Pulteney Practice, Bath
  - Birmingham Clinical Research Centre, Birmingham
  - Stonehill Medical Center, Bolton
  - Avondale Surgery, Chesterfield
  - Chorley Clinical Research Centre, Chorley
  - Saltash Health Center, Cornwall
  - Gomersal Lane Surgery, Dronfield
  - Townhead Research, Irvine
  - Crosby Clinical Research Centre, Liverpool
  - The Symons Medical Center, Maidenhead
  - Manchester Clinical Research Centre, Manchester
  - Greenwood Medical Center, Nottingham
  - Knowle House Surgery, Plymouth
  - Reading Clinical Research Centre, Reading
  - Elm Lane Surgery, Sheffield
  - The Burngreave Surgery, Sheffield
  - Brook Lane Surgery, Southampton
  - St Helier Hospital, Surrey
  - Box Surgery, Wiltshire
  - Bradford Road Medical Center, Wiltshire
  - Eastleigh Surgery, Wiltshire
  - Lovemead Group Practice, Wiltshire
  - Rowden Medical Partnership, Wiltshire
  - St Chad's Surgery, Wiltshire
  - The Health Centre, Wiltshire
  - The Porch Surgery, Wiltshire
  - The Burns Medical Practice, Yorkshire

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First Patient In: 4 October 2005 Last Patient Out: 8 November 2006 A total of 39 investigators at 39 sites in India, Russia, Spain and Denmark received IRB approval to participate in this study and screened and randomized patients.
Pre-assignment Details: Patients with major protocol violations were identified programmatically prior to unblinding to determine who should be excluded from the per protocol population.
Groups:
- Pitavastatin 2 mg QD: Pitavastatin 2 mg daily
- Atorvastatin 10 mg QD: Atorvastatin 10 mg daily
- Pitavastatin 4 mg QD: Pitavastatin 4 mg daily
- Atorvastatin 20 mg QD: Atorvastatin 20 mg daily
Period: Overall Study
Arm/Group | Pitavastatin 2 mg QD | Atorvastatin 10 mg QD | Pitavastatin 4 mg QD | Atorvastatin 20 mg QD
Started | 321 | 103 | 303 | 103
Safety Population | 316 (All randomized patients who received at least one dose of study treatment.) | 102 (All randomized patients who received at least one dose of study treatment.) | 300 (All randomized patients who received at least one dose of study treatment.) | 103 (All randomized patients who received at least one dose of study treatment.)
Completed | 301 | 98 | 288 | 100
Not Completed | 20 | 5 | 15 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pitavastatin 2 mg QD | Atorvastatin 10 mg QD | Pitavastatin 4 mg QD | Atorvastatin 20 mg QD | Total
Number analyzed (Participants) | 316 | 102 | 300 | 103 | 821
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 219 | 75 | 207 | 73 | 574
  >=65 years | 97 | 27 | 93 | 30 | 247
Age Continuous [Mean (Standard Deviation); unit: years] | 58.4 (9.51) | 59.2 (8.63) | 57.9 (10.1) | 58.0 (9.14) | 58.3 (9.58)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 174 | 50 | 164 | 55 | 443
  Male | 142 | 52 | 136 | 48 | 378

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline Low Density Lipoprotein-cholesterol (LDL-C) at Week 12
Time Frame: Baseline to 12 weeks
Population: All patients, irrespective of protocol violations, who had Week 12 measurements, whether on drug or not.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Pitavastatin 2 mg QD | Atorvastatin 10 mg QD | Pitavastatin 4 mg QD | Atorvastatin 20 mg QD
Number analyzed (Participants) | 301 | 98 | 288 | 100
percent change | -37.89 (13.841) | -38.76 (14.582) | -45.5 (14.005) | -43.9 (15.853)

2. Secondary Outcome: Percent Change From Baseline in Total Cholesterol (TC)
Description: Percent change in total cholesterol from baseline to Week 12
Time Frame: Baseline to 12 Weeks
Population: All patients, irrespective of protocol violations, who had Week 12 measurements, whether on drug or not.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Pitavastatin 2 mg QD | Atorvastatin 10 mg QD | Pitavastatin 4 mg QD | Atorvastatin 20 mg QD
Number analyzed (Participants) | 301 | 98 | 288 | 100
percent change | -27.57 (10.359) | -28.92 (11.441) | -33.09 (10.732) | -32.99 (12.073)

3. Secondary Outcome: Percent Change From Baseline in High Density Lipoprotein Cholesterol (HDL-C)
Description: percent change from baseline in high density lipoprotein-cholesterol (HDL-C)
Time Frame: Baseline to 12 weeks
Population: All patients, irrespective of protocol violations, who had Week 12 measurements, whether on drug or not.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Pitavastatin 2 mg QD | Atorvastatin 10 mg QD | Pitavastatin 4 mg QD | Atorvastatin 20 mg QD
Number analyzed (Participants) | 301 | 98 | 288 | 100
percent change | 4.28 (16.501) | 3.42 (16.820) | 4.93 (16.629) | 2.63 (13.803)

4. Secondary Outcome: TC:HDL-C Ratio
Description: Ratio of mean total cholesterol to mean HDL-C at 12 weeks
Time Frame: 12 weeks
Population: All patients, irrespective of protocol violations, who had Week 12 measurements, whether on drug or not.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Pitavastatin 2 mg QD | Atorvastatin 10 mg QD | Pitavastatin 4 mg QD | Atorvastatin 20 mg QD
Number analyzed (Participants) | 301 | 98 | 288 | 100
ratio | 4.018 (1.1294) | 3.763 (0.8667) | 3.583 (1.0961) | 3.79 (1.2052)

5. Secondary Outcome: Triglycerides (TG)
Description: mean triglycerides at 12 weeks
Time Frame: 12 weeks
Population: All patients, irrespective of protocol violations, who had Week 12 measurements, whether on drug or not.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Pitavastatin 2 mg QD | Atorvastatin 10 mg QD | Pitavastatin 4 mg QD | Atorvastatin 20 mg QD
Number analyzed (Participants) | 302 | 98 | 288 | 100
mg/dL | 132.4 (59.82) | 122.2 (57.09) | 124.4 (64.91) | 122.6 (59.01)

6. Secondary Outcome: Non-HDL:HDL Ratio
Description: Ratio of non-HDL to HDL at 12 weeks
Time Frame: 12 weeks
Population: All patients, irrespective of protocol violations, who had Week 12 measurements, whether on drug or not.
Measure: Mean (Standard Deviation)
Arm/Group | Pitavastatin 2 mg QD | Atorvastatin 10 mg QD | Pitavastatin 4 mg QD | Atorvastatin 20 mg QD
Number analyzed (Participants) | 234 | 82 | 250 | 82
Value | 2.993 (1.0935) | 2.770 (0.8846) | 2.601 (1.0961) | 2.710 (1.1771)

7. Secondary Outcome: Apolipoprotein B (Apo B)
Description: Apolipoprotein B at 12 weeks
Time Frame: 12 weeks
Population: All patients, irrespective of protocol violations, who had Week 12 measurements, whether on drug or not.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Pitavastatin 2 mg QD | Atorvastatin 10 mg QD | Pitavastatin 4 mg QD | Atorvastatin 20 mg QD
Number analyzed (Participants) | 295 | 98 | 285 | 99
mg/dL | 114.5 (23.36) | 111.1 (25.12) | 102.3 (22.04) | 102.4 (22.13)

8. Secondary Outcome: Apolipoprotein-A1 (Apo-A1)
Description: Apolipoprotein-A1 at 12 weeks
Time Frame: 12 weeks
Population: All patients, irrespective of protocol violations, who had Week 12 measurements, whether on drug or not.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Pitavastatin 2 mg QD | Atorvastatin 10 mg QD | Pitavastatin 4 mg QD | Atorvastatin 20 mg QD
Number analyzed (Participants) | 295 | 98 | 285 | 99
mg/dL | 164.6 (29.10) | 166 (26.8) | 166.9 (28.01) | 160.9 (26.58)

9. Secondary Outcome: Apo-B:Apo-A1 Ratio
Description: Ratio of Apo-B to Apo-A1 at 12 weeks
Time Frame: 12 weeks
Population: All patients, irrespective of protocol violations, who had Week 12 measurements, whether on drug or not.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Pitavastatin 2 mg QD | Atorvastatin 10 mg QD | Pitavastatin 4 mg QD | Atorvastatin 20 mg QD
Number analyzed (Participants) | 295 | 98 | 285 | 99
ratio | 0.72 (0.228) | 0.68 (0.181) | 0.64 (0.198) | 0.66 (0.205)

10. Secondary Outcome: High Sensitivity C-reactive Protein (Hs-CRP) at 12 Weeks
Description: high sensitivity C-reactive protein (hs-CRP) at 12 weeks
Time Frame: 12 weeks
Population: All patients, irrespective of protocol violations, who had Week 12 measurements, whether on drug or not.
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Pitavastatin 2 mg QD | Atorvastatin 10 mg QD | Pitavastatin 4 mg QD | Atorvastatin 20 mg QD
Number analyzed (Participants) | 301 | 97 | 288 | 100
mg/L | 2.87 (5.101) | 2.39 (3.053) | 3.12 (5.186) | 2.56 (2.958)

11. Secondary Outcome: Oxidized LDL at 12 Weeks
Description: oxidized low density lipoprotein at 12 weeks
Time Frame: 12 weeks
Population: All patients, irrespective of protocol violations, who had Week 12 measurements, whether on drug or not.
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Pitavastatin 2 mg QD | Atorvastatin 10 mg QD | Pitavastatin 4 mg QD | Atorvastatin 20 mg QD
Number analyzed (Participants) | 302 | 98 | 289 | 100
U/L | 59.93 (14.96) | 58.59 (14.679) | 54.32 (13.496) | 54.70 (17.865)

12. Secondary Outcome: National Cholesterol Education Program [NCEP]LDL-C Target Attainment
Description: Number of patients achieving NCEP LDL-C target (LDL-C less than or equal to 130 mg/dL)
Time Frame: up to 12 weeks
Population: All patients, irrespective of protocol violations, who had Week 12 measurements, whether on drug or not.
Measure: Number; unit: Patients
Arm/Group | Pitavastatin 2 mg QD | Atorvastatin 10 mg QD | Pitavastatin 4 mg QD | Atorvastatin 20 mg QD
Number analyzed (Participants) | 315 | 102 | 298 | 102
Patients | 179 | 67 | 232 | 72

ADVERSE EVENTS:
Description: Safety was assessed for all randomized patients who received at least one dose of study drug (Safety Population). The Safety Population contained 821 patients; 616 were treated with pitavastatin and 205 with atorvastatin.
Arm/Group | Pitavastatin 2 mg QD | Atorvastatin 10 mg QD | Pitavastatin 4 mg QD | Atorvastatin 20 mg QD
Serious Adverse Events (participants affected / at risk) | 3/316 | 1/102 | 1/300 | 2/103
Other Adverse Events (participants affected / at risk) | 22/316 | 6/102 | 17/300 | 4/103
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pitavastatin 2 mg QD (N=316) | Atorvastatin 10 mg QD (N=102) | Pitavastatin 4 mg QD (N=300) | Atorvastatin 20 mg QD (N=103)
pruritus generalized (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
acute myocardial infarction (Cardiac disorders) | 1 | 0 | 0 | 0
angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 1
angina unstable (Cardiac disorders) | 0 | 1 | 0 | 0
myocardial infarction (Cardiac disorders) | 0 | 0 | 1 | 0
deafness neurosensory (Ear and labyrinth disorders) | 0 | 0 | 0 | 1
burning sensation (Nervous system disorders) | 1 | 0 | 0 | 0
encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 1
abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pitavastatin 2 mg QD (N=316) | Atorvastatin 10 mg QD (N=102) | Pitavastatin 4 mg QD (N=300) | Atorvastatin 20 mg QD (N=103)
constipation (Gastrointestinal disorders) | 7 | 1 | 3 | 0
nasopharyngitis (Infections and infestations) | 10 | 4 | 8 | 3
myalgia (Musculoskeletal and connective tissue disorders) | 5 | 1 | 6 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days